CLINICAL TRIAL: NCT02376569
Title: An Observational Pilot Study to Characterize Relationships Between Self-reported Information, Game Performance, and Passive Physiology Measures Throughout a Daily Cycle
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-1418
Record Dates: First submitted 2015-01-07; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Energy and Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study intends to collect self-reported information with multiple surveys about lifestyle habits, food and drink, state of mind (happy, sad, etc.) and traits (decision making, general personality, etc.) The purpose of this study is to understand relationships between self-reported information, game performance, and passive physiology measures throughout a daily cycle.

ELIGIBILITY:
Inclusion Criteria:

Must be >=18 years old Must agree to participate via electronic consent Must agree to share e-mail and physical address (final dataset de-identified) Must own a computer and/or smartphone Must be a member of the survey panel and agree to take multiple surveys over 4-6 weeks Must complete the full surveys and not fail attention filters Must be able to access cognition games website and play the games Must be willing to wear a lifestyle assessment sensing device for 1 week

Exclusion Criteria:

Known skin reaction or allergy to metal Known skin reaction or allergy to medical adhesive Participation in another research study, behavior or new drug testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population >=18 years old
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that there are relationships between self-reported information, game performance, and passive physiology measures throughout a daily cycle. | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Marsteller, PhD, Principal Investigator — PepsiCo Global R&D